CLINICAL TRIAL: NCT01053520
Title: Assess the Oral Bioavailability of a New ABT-263 Formulation in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Andrew Krivoshik, MD, PhD, Medical Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: M11-957
Record Dates: First submitted 2009-11-23; First posted 2010-01-21 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Female Subjects
MeSH Terms: interventions — navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence I (Experimental)
  Interventions: Drug: ABT-263
- Sequence II (Experimental)
  Interventions: Drug: ABT-263
- Sequence III (Experimental)
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Period 1: Single (oral) dose of 25 mg of Formulation A Period 2: Single (oral) dose of 25 mg of Formulation B1 Period 3: Single (oral) dose of 25 mg of Formulation B2
  Arms: Sequence I
Drug: ABT-263 — Period 1: Single (oral) dose of 25 mg of Formulation B1 Period 2: Single (oral) dose of 25 mg of Formulation B2 Period 3: Single (oral) dose of 25 mg of Formulation A
  Arms: Sequence II
Drug: ABT-263 — Period 1: Single (oral) dose of 25 mg of Formulation B2 Period 2: Single (oral) dose of 25 mg of Formulation A Period 3: Single (oral) dose of 25 mg of Formulation B1
  Arms: Sequence III

SUMMARY:
This is a Phase 1, randomized, open-label, single center, three period crossover study to determine the oral bioavailability of a new ABT-263 formulation relative to that of the current ABT-263 formulation being administered in ongoing Phase 1/2a studies. Approximately 12 healthy female subjects will be enrolled in this study.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, single center, three period crossover study to determine the oral bioavailability of a new ABT-263 formulation relative to that of the current ABT-263 formulation being administered in ongoing Phase 1/2a studies. Approximately 12 healthy female subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Female and age is between 18 and 55 years, inclusive.
* Must be surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), postmenopausal (for at least 2 years), or practicing at least one acceptable method of birth control.
* Must have negative results for pregnancy tests performed at Screening on a urine sample obtained within 28 days prior to initial study drug administration, and on Period 1 Day -1 on a serum specimen.
* Body Mass Index (BMI) is 18 to 29, inclusive. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Must have adequate bone marrow function per local laboratory reference range (Platelets >/= lower limit of normal range, ANC >/= lower limit of normal range)
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* Must voluntarily sign and date each informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any study-specific procedures.

Exclusion Criteria:

* History of significant sensitivity to any drug
* History of drug or alcohol abuse w/i 6 months or currently receiving Disulfiram
* Known/suspected history of HIV
* History of or active medical condition(s) or surgical procedure(s) that might affect GI motility, pH, absorption
* History of thrombocytopenic associated bleeding w/i 1 year prior to ABT-263
* Significant history of cardiovascular disease (e.g., MI, thrombotic or thromboembolic event in last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, respiratory (except mild asthma), gastrointestinal, hematologic, or hepatic disease or diabetes, cancer, epilepsy, or seizures that in the opinion of the PI would adversely affect her participating in the study.
* Underlying condition predisposing to bleeding or currently exhibits signs of clinically significant bleeding or active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Positive result for drugs of abuse, alcohol, cotinine, hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab).
* Consumed alcohol, grapefruit or starfruit product, or Seville oranges w/i 3 days prior to ABT-263
* Received aspirin, anticoagulation therapy, or any drugs or herbal supplements that affect platelet function w/i 7 days prior to/during ABT-263
* Used any medications, vitamins, or herbal supplements (except contraceptives) w/i 14 days prior to ABT-263
* Received any drug by injection or biologic agent w/i 30 days prior to ABT-263 (except parenteral hormonal contraceptives)
* Used known inhibitors or inducers CYP3A w/i 1 month prior to ABT-263; Received any investigational product w/i 6 weeks prior to ABT-263
* Used tobacco or nicotine-products w/i 6 months prior to ABT-263
* Pregnant or breastfeeding
* Donation or loss of >/=550 mL blood or received transfusion of blood product w/i 8 weeks prior ABT-263
* Currently enrolled in another study.
* The PI decides the subject is unsuitable to receive ABT-263.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Assess the oral bioavailability of Formulation B1 and Formulation B2 via pharmacokinetic measurements relative to Formulation A . | Each formulation assessed via 13 PK timepoints over 4 days

SECONDARY OUTCOMES:
Secondary outcome measures include adverse event monitoring, vital signs, physical examinations, ECGs, and laboratory assessments including pharmacogenetics. | Assessed over the confinement period of 17 days of study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 23602, Waukegan, Illinois, United States